CLINICAL TRIAL: NCT06672484
Title: Gait and Cortical Activity Profile of People With Multiple Sclerosis Presenting With Walking Fatigability
Brief Title: Walking Fatigability and Brain Activity in People With Multiple Sclerosis
Status: Active, not recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: National MS Center Melsbroek (Other); Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Prof. Dr., Hasselt University
Other Study IDs: B1152024000007
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Healthy
Keywords: Multiple sclerosis; walking; fatigue; fatigability; gait; cortical activity; brain activity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: People presenting with multiple sclerosis diagnosis according to the 2017 revisions of the Mcdonald's criteria.
- Healthy people: Inclusion criteria for healthy controls (part A and B): inclusion of age between 18 and 65 years old, sex- and age-matched on a group level.

SUMMARY:
Walking fatigability is a motor impairment happening in approximately 43.5% of people with multiple sclerosis (pwMS). Walking fatigability is defined as a decrease in 10% of distance walked, comparing the first minute with the last minute of the 6-minute walking test (6MWT), which one may call distance walking fatigability. More recently, our research group has found that walking fatigability manifests also in terms of gait quality, with different gait characteristics affected from patient to patient, suggesting that different gait profiles might be observed for walking fatigability. One possible explanation for the walking fatigability motor impairment is the lower capacity or neural reserve of pwMS to sustain optimal levels of cortical activity to either maintain performance (i.e., distance walked) or gait quality.

The study proposes two research questions. Both part A and B are observational studies.

The study includes 70 pwMS and 30 healthy controls. The study consists of 3 tests. The clinical assessment session will be composed of responses to different questionnaires, while parts A and B comprehend walking overground (part A) or on fixed-speed treadmill (part B).

Part A Session 1 (1 hour and 30minutes, including equipment preparation and rest time).

First, anthropometric characteristics and measurements of force, spasticity, cognition, walking speed, and performance foot tap test will be performed. For cortical activity measurement of the prefrontal cortex, supplementary motor area, premotor cortex, and primary motor cortex, a functional Nears-infrared Spectroscopy (fNIRS) will be positioned in the participant's head. Wearable sensors will be positioned in a pre-defined body position for the measurement of gait characteristics. Both gait characteristics and cortical brain activation will be measured concomitantly during fast and comfortable speed short walking (10 trials of 15 seconds with 25-30 seconds standing still resting periods between trials, in a block design) before and after and during a prolonged walking (6-minute walking test (6MWT)) protocols. A resting period of 20 minutes will be provided to the participants before the beginning of the 6MWT.

Part B. Participants who participated in Part A will be invited to participate in Part B. This study also consists of a single visit that is 1 hour and 30 minutes long (preparation and assessment included). The participants will be asked to walk on an immersive treadmill in two fixed-speed conditions (relative to 80% and 50% of the Timed 25-foot Walking test) while infrared cameras will record the reflective markers position. Forty minutes of rest will be provided to the participants between the fixed-speed conditions.

DETAILED DESCRIPTION:
Methodology Recruitment strategy. Participants will be recruited from the Flemish MS rehabilitation centers Melsbroek (NMSC) and Overpelt (Noorderhart RMSC), as well as the REVAL research center inUHasselt. Information flyers will be distributed in the centers and via information placed on the website and social media of REVAL and the Flemish MS society. We will search age and sex-matching subjects for the healthy controls, considering a 5-year range per subject.

After giving informed consent, demographics of age and gender, as well as MS-related information such as EDSS, type of MS, and years since diagnosis, will be collected and provided by the centers or via self-report. The participants will be instructed to keep their normal routine and avoid extraneous physical activity at least 24 hours before the data collection session.

Experiment outline. The study proposes two research questions and will be performed in three days. The first day is the clinical assessment/screening of the participants (common for Part A and B). Part A is an observational study (2nd day), and Part B is an observational and feasibility study (3rd day).

Clinical assessment/screening The participants will be contacted to verify their interest and eligibility (inclusion and exclusion criteria) to participate in the study. In the case of inclusion in the study, different questionnaires will be sent to the participants to fill in: Falls Efficacy Scale International (FES-I) for fear of falling, Multiple Sclerosis Walking Scales (MSWS-12) and 10 questions encompassing gait items for walking perceived ability [11], Pittsburgh Fatigability Scale (PFS) for perceived fatigability, Modified Fatigue Impact Scale (MFIS) for perceived fatigue, the Brief Pain Inventory (BPI, short form) for the assessment of perceived pain, Multiple Sclerosis Spasticity Scale 88 (MSWS-88, section 5 and 6) to verify the impact of spasticity in the walking and movement ability and Brief Self-Control Scale (BSCS) for self-control evaluation. Specifically for the pwMS, the Patients Disease Determined Steps (PDDS) will be asked in order to know the self-perceived level of disability. Participants will also be asked and oriented to measure their head's circumference for the functional near-infrared spectroscopy (fNIRS) measurement. In case the patient is contacted in the MS centers (MS Rehabilitation Center- Pelt and National MS Center Melsbroek), the therapist will provide the questionnaires, measure the head size of the participants, and obtain the level of disability (measured by the expanded disability status scale- EDSS). The skin color, type, and color of the hair will be noted to assist in the fNIRS analysis.

Part A- Assessment The study includes 70 pwMS and 30 healthy controls. The study consists of a single visit (1 hour and 30 minutes duration, including equipment preparation and rest periods). Participants will be asked to wear shorts or legging pants for better fixation of the sensors. Anthropometric characteristics such as age, weight, height, and sex will be asked and measured. Moreover, for pwMS, the time from the diagnosis, MS phenotype, and medications that could influence fatigue or walking performance will also be recorded. The symbol digit modalities test (SDMT) will evaluate the cognitive processing speed. Afterward, the modified Ashworth scale (MAS) will be used to check the muscle spasticity of the knee flexors/extensors and ankle flexors/extensors. The motricity index will be performed for muscle strength measurement, followed by the performance of the timed 25-foot walking test (T25FWT). For cortical activity measurement of the prefrontal cortex, supplementary motor area, premotor cortex, and primary motor cortex, a fNIRS will be positioned in the participants head. Wearable sensors will be positioned in a pre-defined body position to measure gait characteristics. Both gait characteristics and cortical brain activation will be measured concomitantly during short walking (10 trials of 15 seconds with 25-30 seconds standing still resting periods between trials, in a block design) before and after and during a prolonged walking (6-minute walking test (6MWT)) protocols. Before the beginning of the 6MWT, two questions will be asked to the participants: "Do you slow down when walking for a while?" and "Do you feel a worsening of your smoothness when walking for a while?" where they will have to rate between 1 ("not at all") and 5 ("Extremely"). A questionnaire about their perceived gait quality changes, comparing the end with the beginning of the 6MWT, will be asked through the Perception of Gait Quality Change (PGQC).

Part B- Assessment The study includes 30 pwMS and 30 healthy controls. Participants who participated in Part A will be invited to participate in Part B. Participants will be asked to wear shorts or legging pants for better fixation of the sensors and the reflective markers. This study also consists of a single visit of 1 hour and 30 minutes (preparation and assessment included). The wearable sensors will be positioned in the participants following the same setup as part A. Reflective markers will be positioned in body landmarks. The participants will be asked to walk on an immersive treadmill in two fixed-speed conditions (relative to 80% and 50% of the T25FW), while infrared cameras will record the reflective markers position. The participants will also be asked about previous experience walking on a treadmill.

PART A. ASSESSMENT. Outcome measures specifications Foot tap test. The participants will have to perform a foot tap test as fast and with higher amplitude as possible for 6 times: i) 2 times 10 seconds for each foot, with resting period of 1 minute between the trials and ii) one time, each foot, for 1 minute. The two times 10 seconds for each foot will be repeated after the short walking test after the 6MWT. Inertial measurement units will be position on the top of their feet for frequency and amplitude of the movement measurement concomitantly with the record of cortical brain activity measurement. A baseline period of 15 seconds, preceding each trial, will be performed for the cortical brain activity.

Short walking test. The participants will be instructed to walk at their maximum (5 times) and comfortable speed (5 times) in blocks of 15 seconds, with rest periods ranging from 25 to 30 seconds before and after the 6MWT. The order of the first four trials will be consistent among participants (starting with 2 fast walking followed by 2 comfortable walking). The remaining of the trials will be randomized. The different resting periods were chosen to prevent the participants from anticipating the beginning of the trial, minimizing the effects of anticipation on cortical brain activation. During the resting periods, the participants will be instructed to perform a simple cognitive task of counting down starting from 50 to prevent mind wandering. The software Psychophy will be used to draw the experimental procedure and synchronize the wearable sensors and fNIRS equipment. Standardized audio instructions will be provided to the participants on what they will have to do and the countdown for the beginning of the task.

Walking capacity and fatigability test. Participants will perform the 6MWT. During the 6MWT, participants will be instructed to safely walk as fast as possible to cover a maximal individual distance for 6 min on a 25m walkway with turns at both ends. No verbal encouragement will be provided to the participants and every minute completed of the test will be informed by the research staff. Patients will be allowed to use an assistive device if needed, and no rest during the 6MWT will be allowed.

Measuring gait:

Participants will be equipped with 10 wearable sensors (OPAL V.2, APDM, USA, https://www.apdm.com/wearable-sensors/) to measure gait characteristics in different gait domains. Two sensors will be strapped on their feet, two on each tibia, two on each thigh, two on each wrist, one on their lumbar (L4), and one on the sternum.

Measuring cortical brain activity:

The measurement of cortical brain activity will follow the guidelines to assess gait and posture using fNIRS . Participants will wear a portable fNIRS cap with a backpack containing the fNIRS device on the back. The size of the cap will change in accordance with the head size of each participant. The fNIRS system is composed of 16 sensors and 16 detectors and will be positioned in the cap to measure the following regions of interest: the prefrontal cortex (Broadman area 9, 10, and 46), supplementary motor area (Broadman area 6), premotor cortex (Broadman area 6), and primary motor cortex (Broadman area 4). These areas correspond to the areas involved in the brain's human control for walking.

PART B. ASSESSMENT. Outcome measures specifications 6-minute walking test (6MWT) fixed speed. The participants will perform the 6MWT in a two-belt treadmill, with two force platforms embedded, in the Gait Real-Time interactive laboratory (GRAIL), in two fixed speed conditions: i) 80% of the walking speed obtained in the T25FW and ii) 50% of the walking speed obtained in the T25FW. The order of the fixed-speed treadmill conditions will be randomized and counterbalanced between groups. Forty minutes will be provided to the participants between the fixed-speed conditions. The GRAIL (Motekforce Link, Amsterdam, the Netherlands) will assess gait characteristics changes over the fixed-speed 6MWT. This system allows real-time recording of body movement in a high-resolution recording by means of a 3D motion capture system (10 cameras Vicon Motion System® with a data collection frequency set at 100 Hz). Twenty-two passive reflective markers (HBM lower body model) will be positioned on the bony landmarks of participants.

ELIGIBILITY:
Inclusion Criteria (part A and B):

* age between 18 and 65 years old
* a diagnosis of MS (2017 revisions of the McDonalds criteria) with EDSS 1 up to 6.5 (part A) and with EDSS 1 up to 5.5 (part B) OR minimal punctuation of 2 in the MSWS-12 for one of the items: 7, 10, 11, and 12 (for pwMS)
* no relapses 1 month preceding the start of the study (for pwMS)
* ability to walk for 6 minutes without rest

Exclusion Criteria (Part A and B):

* Cognitive impairment hindering understanding of study instructions,
* Pregnancy
* Musculoskeletal disorders in the lower limbs that are not related to MS.
* PwMS needing an assistive device to walk can not be included in part B given safety reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Flemish MS rehabilitation centers Melsbroek (NMSC) and Overpelt (Noorderhart RMSC), as well as the REVAL research center in UHasselt. Information flyers will be distributed in the centers and via information placed on the website and social media of REVAL and the Flemish MS society. We will search age and sex-matching subjects for the healthy controls, considering a 5-year range per subject.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (hip, knee and ankle joints) during the gait cycle | Day 2 and day 3
  The angle of the hip, knee, and ankle joints in the sagittal (flexion-extension), coronal (adduction-abduction), and transversal (rotation) plans during the gait cycle
Toe-Off angle | Day 2 and day 3
  The plantar flexion of the foot in the last moment of contact of the feet with the floor
Foot Strike angle | Day 2 and day 3
  The dorsiflexion of the feet in the heel strike
Relative concentration of oxyhemoglobin and deoxyhemoglobin | Day 2
  The cortical brain activation will be obtained through functional near-infrared spectroscopy (fNIRS). The fNIRS measures the relative concentration of oxyhemoglobin and deoxyhemoglobin in the brain tissue, more specifically, in the brain cortex. The following brain regions will be measured:
  * Frontopolar cortex (Broadman area 10)
  * Dorsolateral prefrontal cortex (Broadman 9 and 46)
  * Primary motor cortex (Broadman area 4)
  * Supplementary motor area (Broadman area 6)
  * Premotor cortex (Broadman area 6)
Gait Speed | Day 2 and day 3
  The anteroposterior distance, divided by the gait cycle duration (two subsequent heel strikes of the same leg).
Cadence | Day 2 and day 3
  Number of steps made per minute (both legs)
Step Duration | Day 2 and day 3
  The duration from the heel strike of a leg with the heel strike of the contralateral leg
Step Duration variability | Day 2 and day 3
  The coefficient of variation calculated from the step duration variable
Ground reaction force | Day 3
  It is the amount of force produced against the floor by a person. It will measured in the three directions: vertical, anteroposterior, and medial-lateral.
Fatigability index | Day 2 and day 3
  A fatigability index will be applied for all gait parameters for the 6-minute walking test and the treadmill walking listed in accordance with the following sentence:
  fatigability index: ((gait parameters at minute n- gait parameter at minute 1)/gait parameter at minute 1)*100.
Perception of gait quality change (PGQC) | Day 2 and day 3
  It is a questionnaire to measure the capacity of the person to perceive changes in his/her gait after walking for a prolonged time. Here, this questionnaire is asked after the 6-minute walking test (6MWT). The questionnaire is in a Likert-type score, ranging from -3 (very much worse) to 3 (very much improved).
Distance walked index (DWI) | Day 2
  The distance walked index (DWI) will be applied to the distance walked in each minute of the 6-minute walking test using the following formula:
  DWI(%) = ((distance walked at minute n- distance walked at minute 1)/ distance walked at minute 1)*100
6-minutes walking test | Day 2
  The total distance and the distance walked, in meters, minute-by-minute will be recorded during the 6-minutes walking test.

SECONDARY OUTCOMES:
Joint power during the gait cycle | Day 3
  Joint power represents the overall rate, amount, and timing of energy generated and dissipated by all the muscles and ligaments surrounding a joint. It will be calculated specifically for the hip, knee and ankle joints during the gait cycle. It specifically uses data from kinematic and kinetic for it calculation.
Momentum | Day 3
  It is the quantity of motion the body has while walking, calculated as mass times velocity, helping to maintain forward movement. It will be calculated for hip, knee and ankle joints during the gait cycle.
Falls Efficacy Scale International (FES-I) | Day 1
  A questionnaire assessing fear of falling. It includes 16 items, with scores ranging from 16 to 64, where higher scores indicate greater fear of falling.
Multiple Sclerosis Walking Scale (MSWS-12) | Day 1
  A 12-item self-reported questionnaire measuring the impact of MS on walking. Scores range from 12 to 60, with higher scores indicating greater walking impairment
Pittsburgh Fatigability Scale (PFS) | Day 1
  A 10-item scale measuring perceived physical and mental fatigability from activities of daily living. The total score ranges from 0 to 50, where higher scores indicate greater fatigability.
Modified Fatigue Impact Scale (MFIS) | Day 1
  A 21-item questionnaire assessing the impact of fatigue on physical, cognitive, and psychosocial functioning. Scores can be obtained separately or in total (physical: 0-36; cognitive: 0-40; psychosocial: 0-8; total: 0-80). Higher scores reflect a greater impact of fatigue.
Brief Self-Control Scale (BSCS) | Day 1
  A 13-item questionnaire evaluating self-regulation abilities. Scores range from 13 to 65, with higher scores indicating better self-control.
Multiple Sclerosis Spasticity Scale-88 (MSSS-88) | Day 1
  An 88-item questionnaire measuring spasticity and its effect on daily functioning in MS. In this study, we used sections 5 and 6 only as they reflect daily living activities. Higher scores indicating greater spasticity
Brief Pain Inventory (BPI, short form) | Day 1
  A 16-item questionnaire assessing pain severity and interference with daily life. Pain severity scores range from 0 to 10, and interference scores from 0 to 70, with higher scores indicating more severe pain and greater impact on daily activities.
Expanded Disability Status Scale (EDSS) | Day 1
  It is a classification rate of disability for people with multiple sclerosis ranging from 0 (no disability) to 10 (bedridden due to MS).
Modified Ashworth Scale (MAS) | Day 2
  It measures muscle spasticity in the muscles. Here, the spasticity in the lower limb muscles of the three joints (knee, hip and ankle) will be measured.
Motricity index (MI) | Day 2
  It is a clinical test to measure the motor function/muscle strength of lower and upper limb muscles. In this study, the muscle strength of the hip flexors, knee extensors, and ankle dorsiflexion will be measured.
Borg scale | Day 2 and day 3
  It is a scale to identify how much exertion a person is doing at that time point. It ranges from 0 ("No exertion at all") to 10 ("Maximal effort"). The Borg will be asked before and after the 6-minute walking test, as well as the two conditions of treadmill walking.
Variability interpeak (Foot tap test) | Day 2
  The variability of the duration between each foot tap performed.
Number of foot tap (Foot tap test) | Day 2
  The amount of foot tap performed.
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Day 1
  A 20-item questionnaire assessing how fatigue impact on quality of life. Fatigue severity scores range from 1 (Does not apply at all) to 5 (Applies completely), with higher scores indicating more severe fatigue and greater impact on daily activities.

OTHER OUTCOMES:
Lyapunov Exponent | Day 2
  Measure to what extent two trajectories diverge over time (i.e., acceleration)
Double Support | Day 2 and day 3
  The percentage of the gait cycle in which both feet are in contact with the floor
Patients determined disease steps (PDDS) | Day 1
  It is a self-reported scale used by individuals with multiple sclerosis (MS) to rate their level of disability. It ranges from 0 (normal) to 8 (bedridden), focusing primarily on mobility and walking ability.
Timed 25-foot walking test (T25FW) | Day 2
  It is a walking capacity test where the person has to walk as fast as possible, without running, for 7.62 meters. The time needed to complete is recorded in two valid trials.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - University of Hasselt, Diepenbeek, Limburg
  - National MS Melsbroek, Melsbroek
  - Noorderhart Rehabilitation & MS centre, Overpelt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santinelli FB, Abasiyanik Z, Dalgas U, Ozakbas S, Severijns D, Gebara B, Maamagi H, Romberg A, Rasova K, Santoyo-Medina C, Ramari C, Leone C, Feys P. Prevalence of distance walking fatigability in multiple sclerosis according to MS phenotype, disability severity and walking speed. Ann Phys Rehabil Med. 2025 Feb;68(1):101887. doi: 10.1016/j.rehab.2024.101887. Epub 2024 Dec 9. No abstract available. PMID 39657457
- [Background] Van Geel F, Veldkamp R, Severijns D, Dalgas U, Feys P. Day-to-day reliability, agreement and discriminative validity of measuring walking-related performance fatigability in persons with multiple sclerosis. Mult Scler. 2020 Nov;26(13):1785-1789. doi: 10.1177/1352458519872465. Epub 2019 Sep 9. PMID 31496362
- [Background] Van Geel F, Hvid LG, Van Noten P, Eijnde BO, Dalgas U, Feys P. Is maximal muscle strength and fatigability of three lower limb muscle groups associated with walking capacity and fatigability in multiple sclerosis? An exploratory study. Mult Scler Relat Disord. 2021 May;50:102841. doi: 10.1016/j.msard.2021.102841. Epub 2021 Feb 10. PMID 33621946
- [Background] Strzok S, Cleanthous S, Pompilus F, Cano SJ, Marquis P, Cohan S, Goldman MD, Kresa-Reahl K, Petrillo J, Castrillo-Viguera C, Cadavid D, Chen SY. Development of a gait module to complement the 12-item Multiple Sclerosis Walking Scale: a mixed methods study. Mult Scler J Exp Transl Clin. 2018 Jun 26;4(2):2055217318783766. doi: 10.1177/2055217318783766. eCollection 2018 Apr-Jun. PMID 30090638
- [Background] Sehle A, Mundermann A, Starrost K, Sailer S, Becher I, Dettmers C, Vieten M. Objective assessment of motor fatigue in Multiple Sclerosis using kinematic gait analysis: a pilot study. J Neuroeng Rehabil. 2011 Oct 26;8:59. doi: 10.1186/1743-0003-8-59. PMID 22029427
- [Background] Sato S, Lim J, Miehm JD, Buonaccorsi J, Rajala C, Khalighinejad F, Ionete C, Kent JA, van Emmerik REA. Rapid foot-tapping but not hand-tapping ability is different between relapsing-remitting and progressive multiple sclerosis. Mult Scler Relat Disord. 2020 Jun;41:102031. doi: 10.1016/j.msard.2020.102031. Epub 2020 Feb 27. PMID 32172213
- [Background] Santinelli FB, Ramari C, Poncelet M, Severijns D, Kos D, Pau M, Kalron A, Meyns P, Feys P. Between-Day Reliability of the Gait Characteristics and Their Changes During the 6-Minute Walking Test in People With Multiple Sclerosis. Neurorehabil Neural Repair. 2024 Feb;38(2):75-86. doi: 10.1177/15459683231222412. Epub 2024 Jan 16. PMID 38229519
- [Background] Nagels-Coune L, Benitez-Andonegui A, Reuter N, Luhrs M, Goebel R, De Weerd P, Riecke L, Sorger B. Brain-Based Binary Communication Using Spatiotemporal Features of fNIRS Responses. Front Hum Neurosci. 2020 Apr 15;14:113. doi: 10.3389/fnhum.2020.00113. eCollection 2020. PMID 32351371
- [Background] Menant JC, Maidan I, Alcock L, Al-Yahya E, Cerasa A, Clark DJ, de Bruin ED, Fraser S, Gramigna V, Hamacher D, Herold F, Holtzer R, Izzetoglu M, Lim S, Pantall A, Pelicioni P, Peters S, Rosso AL, St George R, Stuart S, Vasta R, Vitorio R, Mirelman A. A consensus guide to using functional near-infrared spectroscopy in posture and gait research. Gait Posture. 2020 Oct;82:254-265. doi: 10.1016/j.gaitpost.2020.09.012. Epub 2020 Sep 18. PMID 32987345
- [Background] Leone C, Severijns D, Dolezalova V, Baert I, Dalgas U, Romberg A, Bethoux F, Gebara B, Santoyo Medina C, Maamagi H, Rasova K, Maertens de Noordhout B, Knuts K, Skjerbaek A, Jensen E, Wagner JM, Feys P. Prevalence of Walking-Related Motor Fatigue in Persons With Multiple Sclerosis: Decline in Walking Distance Induced by the 6-Minute Walk Test. Neurorehabil Neural Repair. 2016 May;30(4):373-83. doi: 10.1177/1545968315597070. Epub 2015 Jul 27. PMID 26216790
- [Background] Herold F, Wiegel P, Scholkmann F, Thiers A, Hamacher D, Schega L. Functional near-infrared spectroscopy in movement science: a systematic review on cortical activity in postural and walking tasks. Neurophotonics. 2017 Oct;4(4):041403. doi: 10.1117/1.NPh.4.4.041403. Epub 2017 Aug 1. PMID 28924563
- [Background] Goldman MD, Chen S, Motl R, Pearsall R, Oh U, Brenton JN. Progression risk stratification with six-minute walk gait speed trajectory in multiple sclerosis. Front Neurol. 2023 Oct 4;14:1259413. doi: 10.3389/fneur.2023.1259413. eCollection 2023. PMID 37859654
- [Background] Filli L, Sutter T, Easthope CS, Killeen T, Meyer C, Reuter K, Lorincz L, Bolliger M, Weller M, Curt A, Straumann D, Linnebank M, Zorner B. Profiling walking dysfunction in multiple sclerosis: characterisation, classification and progression over time. Sci Rep. 2018 Mar 21;8(1):4984. doi: 10.1038/s41598-018-22676-0. PMID 29563533
- [Background] Baert I, Freeman J, Smedal T, Dalgas U, Romberg A, Kalron A, Conyers H, Elorriaga I, Gebara B, Gumse J, Heric A, Jensen E, Jones K, Knuts K, Maertens de Noordhout B, Martic A, Normann B, Eijnde BO, Rasova K, Santoyo Medina C, Truyens V, Wens I, Feys P. Responsiveness and clinically meaningful improvement, according to disability level, of five walking measures after rehabilitation in multiple sclerosis: a European multicenter study. Neurorehabil Neural Repair. 2014 Sep;28(7):621-31. doi: 10.1177/1545968314521010. Epub 2014 Feb 6. PMID 24503204